CLINICAL TRIAL: NCT05718973
Title: Efficacy of a Short, Animated Storytelling Video to Boost Psychological Capital in the Post-pandemic Era: a Randomized Controlled Trial
Brief Title: A Short, Animated Storytelling Video to Boost Psychological Capital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: Stanford University (Other); Heidelberg University (Other)
Responsible Party: Principal Investigator, PD Dr. Alexander Supady, Attending Physician, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EduEntertainPsy_23
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Psychological Capital
Keywords: psychological capital; education entertainment intervention; short, animated storytelling

STUDY DESIGN:
Intervention Model Description: This is a 4-armed, parallel, randomized controlled trial, conducted purely online
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All study investigators and researchers involved in the data analyses will remain blinded to the trial arm allocation for the entire study duration. Unblinding will not be required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Arm (Experimental): At Time 1, the Intervention Arm will view a short, animated storytelling video designed to promote psychological capital and, immediately thereafter, complete the CPC-12R, the GQ-6 as well as a single-item validated happiness scale.
  Two weeks later, the participants will complete the CPC-12R, the GQ-6 and the single-item validated happiness scale.
  Interventions: Other: short, animated storytelling video (intervention video)
- Scale-Exposed Control Arm (No Intervention): The Scale-Exposed Control Arm will watch no video content at Time 1, but will complete the CPC-12R, the GQ-6 as well as a single-item validated happiness scale.
  Two weeks later, the participants will complete the CPC-12R, the GQ-6 and the single-item validated happiness scale.
- Attention Placebo Control Arm (Placebo Comparator): The Attention Placebo Control Arm will view an attention placebo control video, unrelated to the outcomes measured in this trial, before completing the CPC-12R, the GQ-6 and the single-item validated happiness scale.
  Two weeks later, the participants will complete the CPC-12R, the GQ-6 and the single-item validated happiness scale.
  Interventions: Other: short, animated storytelling attention placebo video
- Un-exposed Control Arm (No Intervention): The Un-exposed Control Arm will neither watch video content, nor complete the CPC-12R, the GQ-6 and the single-item validated happiness scale at Time 1.
  Two weeks later, the participants will complete the CPC-12R, the GQ-6 and the single-item validated happiness scale.

INTERVENTIONS:
Other: short, animated storytelling video (intervention video) — Participants in the Intervention Arm will view a short, animated storytelling video designed to promote psychological capital.
  Arms: Intervention Arm
Other: short, animated storytelling attention placebo video — The Attention Placebo Control Arm will view an attention placebo control video, unrelated to the outcomes measured in this trial.
  Arms: Attention Placebo Control Arm

SUMMARY:
This study will evaluate the effect of a short, animated storytelling intervention video on positive psychological capital intervention on immediate and medium-term psychological capital and related constructs, gratitude and happiness. We will also measure voluntary engagement with the content of the short, animated storytelling intervention video on positive psychological capital.

In this 4-armed, parallel, randomized controlled trial, 10,000 adult, US participants will be randomly assigned to (1) a short, animated storytelling intervention video on positive psychological capital followed by the psychological capital , gratitude and happiness surveys (2) the surveys only, (3) an attention placebo control video followed by the before mentioned surveys, and (4) an arm that is exposed to neither the video nor the surveys. Two weeks later, participants in all four arms will complete all of the surveys.

The primary outcome is psychological capital (immediate and medium-term). Secondary outcomes are gratitude and happiness (immediate and medium-term) as well as voluntary engagement with the short, animated storytelling video content.

ELIGIBILITY:
Inclusion Criteria:

* Registration with the Prolific platform

Exclusion Criteria:

* none

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10000 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Immediate effect of the short, animated storytelling intervention video on positive psychological capital | immediately after watching the video
  The immediate effect of the short, animated storytelling intervention video on positive psychological capital, as measured by the CPC-12R, the GQ-6 and the single-item validated happiness scale.

SECONDARY OUTCOMES:
Medium-term effect of the short, animated storytelling intervention video on psychological capital | 2 weeks
  The medium-term effect of the short, animated storytelling intervention video on psychological capital after two weeks.
Immediate effect of the short, animated storytellingintervention video on gratitude and happiness | immediately after watching the video
  The effect of the short, animated storytellingintervention video on gratitude and happiness, both related to the construct of positive psychological capital
Medium-term effect of exposure to psychological capital and related psychological scales on these same outcomes | 2 weeks
  The effect of exposure to psychological capital and related psychological scales on these same outcomes, measured two weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Till Bärnighausen, Prof. Dr., Principal Investigator — Heidelberg University

IPD SHARING:
Plan to Share IPD: No
Currently not planned. Individual requests may be directed to the corresponding author.

REFERENCES:
- [Derived] Adam M, Rohr J, Greuel M, Nguyen K, Aziz MAE, Gates J, Uberreiter C, Supady A, Barnighausen T. Measuring the effect of short, animated storytelling videos to boost psychological capital in US adults: a randomized controlled trial. Sci Rep. 2025 Nov 18;15(1):40326. doi: 10.1038/s41598-025-26894-1. PMID 41254108